CLINICAL TRIAL: NCT01784393
Title: Chemoradiation With Capecitabine for Palliation of Pain From Bone Metastasis
Brief Title: Chemoradiation for Bone Metastasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bone-X-11
Record Dates: First submitted 2013-01-14; First posted 2013-02-05 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2007-04

CONDITIONS: Breast Cancer; Bone Metastasis; Pain
MeSH Terms: conditions — Breast Neoplasms; Pain | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: chemoradiation

SUMMARY:
Pain from bone metastases of breast cancer origin is treated with localized radiation. Modulating doses and schedules has shown little efficacy in improving results. Given the synergistic therapeutic effect reported for combined systemic chemotherapy with local radiation in anal, rectal, and head and neck malignancies, the investigators sought to evaluate the tolerability and efficacy of combined capecitabine and radiation for palliation of pain due to bone metastases from breast cancer Hypothesis: Given the hypothesis that regimens employing greater intensity radiation yield higher rates of pain relief, radiosensitization using a tumor targeted drug like Xeloda should improve the rate of complete pain relief as compared to radiosensitization with 5FU alone.

Primary Objective:

To determine the frequency and duration of pain relief and narcotic relief for the proposed regimen.

Secondary Objective:

To determine the toxicity of concurrent Capecitabine and radiotherapy in breast cancer patients with bone metastases.

DETAILED DESCRIPTION:
BACKGROUND

Much of the clinical practice of oncology involves palliative care. In this setting ,the emphasis is on alleviation of symptoms and preservation or improvement of quality of life. A large body of clinical evidence documents the effectiveness of local-field external beam radiotherapy in palliation of pain from osseous metastases (1). Despite this general agreement, controversy remains regarding the optimal dose and fractionation schedule. Prospective phase III clinical trials (2-6), today, have failed to demonstrate superiority of one schedule over another ,and as a result, the patterns of practice of remain diverse in duration and intensity.

Between 1974 and 1980 the RTOG conducted a large national study to determine the effectiveness of five different dose fractionation schedules(2). A total of 1016 patients were entered ,266 into a "solitary metastasis" stratum, and 750 into a "multiple metastasis " stratum. The former were randomly assigned to treatment with 40,5Gy in 15 fractions or 20Gy in 5 fractions. The latter were assigned to 30Gy in 10 fractions, 15 Gy in5 fractions ,20 Gy in 5 fractions, or 25 Gy in 5 fractions. A quantitative measure of pain ,based on severity and frequency of pain, and the type and frequency of pain medications used, was devised to evaluate response. Overall, 89% of patients experienced minimal relief. There were no significant difference between the treatment arms in both strata. The initial pain score was found to be a useful predictor ; patients with high score were less likely to respond and were less likely to experience a complete response. Patients with breast and prostate cancer were significantly more likely to respond than patients with lung or other primary lesions. Patients completing their treatment as planned had significantly higher rates of complete response than those who did not .While some relief was experienced almost invariably within the first four weeks, complete relief was first reported later than four weeks after start of treatment in about 50 % of patients .The median duration of minimal and complete pain relief was 20 and 12 weeks ,respectively. There were no significant differences in duration of pain relief between the different arms It was concluded that all treatment dose schedules were equally effective.

A reanalysis of the RTOG study was reported by Blitzer (7).Using a stepwise logistic regression, he examined the effect of the number of fractions, the dose per fraction, and solitary versus multiple metastases, on the probability of attaining complete pain relief and the need for retreatment. This multivariate technique allowed patients with solitary and multiple metastases to be analyzed together. By increasing the number of subjects and events the statistical power of the analysis was outcome. There was no correlation of the time dose factor with outcome (8). It was concluded that the more protracted schedules resulted in improved pain relief.

Price et al. randomized 288 patients to receive either 8 Gy in one fraction or 30 Gy in 10 daily fractions. Pain was assessed using a questionnaire completed by the patients at the home on a daily basis. No differences were found in the probability of attaining pain relief, the speed of onset or the duration of relief between the two arms(4). Hoskin et al. randomized 270 patients to receive either 4 Gy or 8 Gy in one fraction (3) Pain assessed by the patient) and analgesic usage were recorded before treatment and at 2,4,8 and 12 weeks. At 4 weeks the response rates were 69% for 8 Gy and 44% for 4 Gy (p<0.001). The duration of the effect was independent of dose.

Two other randomized trials have been reported (5,6). Given the small difference in the Biological Effective Dose ( BED) between the arms (6) and the small number of patients accrued (5,6), it is not surprising that no differences between the treatment arms were detected.

RTOG have reported the results of a pooled data dose response analysis (11). A computerized literature search was conducted to identify prospectively randomized clinical studies which addressed this issue and the results of these studies (2 6) were pooled together to form a database for analysis. The endpoint selected for analysis was complete response (CR). It was felt that this endpoint was most likely to be evaluated in a consistent fashion by different investigators. One study (6) was excluded from the analysis because outcome was not reported using conventional definitions of complete and partial response. To allow comparison of the different study arms, the BED was calculated for each schedule. Odds ratios calculated for various dose levels showed a statistically significant increase from 1.00 to 3.32 as the BED increased from 14.4 Gy to 5 1.4 Gy.

For the first time, RTOG analysis demonstrated a highly significant dose response relationship for palliation of pain from bone metastases with radiotherapy. Furthermore, there was no evidence of flattening of the dose¬-response curve within the dose range tested, suggesting that further gains can be realized at doses outside of the range tested. We propose a phase II clinical trial in which the biological effective dose will be increased by the concurrent use of a radiosensitizer. The main advantage of this approach over escalation of the physical dose is the avoidance of increase in the overall treatment time.

Capecitabine is a fluoropyrimidine carbamate with antineoplastic activity. It is an orally administered systemic prodrug of 5' deoxy 5 fluorouridine (5' DFUR) which is converted to 5 Capecitabine is readily absorbed from the gastrointestinal tract. In the liver, a 60 kDa carboxyesterase hydrolyzes much of the compound to 5' deoxy 5 fluorocytidine (5' DFCR). Cytidine deaminase, an enzyme found in most tissues, including tumors, subsequently converts 5' DFCR to 5' deoxy 5 fluorouridine (5' DFUR).. The enzyme, thymidine phosphorylase (dThdPase), then hydrolyzes 5' DFUR to the active drug 5 FU. Many tissues throughout the body express thymidine phosphorylase. Some human carcinomas express this enzyme in higher concentrations than surrounding normal tissues. Both normal and tumor cells metabolize 5 FU to 5¬fluoro 2 deoxyuridine monophosphate (FdUMP) and 5 fluorouridine triphosphate (FUTP). These metabolites cause cell injury by two different mechanisms. First, HUMP and the folate cofactor, N5 10¬methylenetetrahydrofolate, bind to thymidylate synthase (TS) to form a covalently bound ternary complex. This binding inhibits the formation of thymidylate from uracil. Thymidylate is the necessary precursor of thymidine triphosphate, which is essential for the synthesis of DNA, so that a deficiency of this compound can inhibit cell division. Second, nuclear transcriptional enzymes can mistakenly incorporate FUTP in place of uridine triphosphate (UTP) during the synthesis of RNA. This metabolic error can interfere with RNA processing and protein synthesis. Capecitabine is already approved for use in patients with metastatic breast cancer resistant to both paclitaxel and an anthracycline containing chemotherapy regimen.

Although 5FU is an established radiosensitizer, the exact mechanism by which it enhances cell kill is not well understood. Sensitization is schedule dependent and is maximal when a cytocidal concentration of 5FU is given after the radiation exposure (12). The effect does not result from increased sublethal damage or inhibition of sublethal damage repair (12,13). Current evidence suggests that radiosensitization by 5FU is mediated through its effects on DNA rather then RNA (14). In vivo (15) as well as clinical studies (16) have demonstrated the superiority of continuous over bolus infusion of 5FU.

Over the last several decades, concurrent 5FU and radiation have been used successfully in a variety of malignancies. Several important lessons have been learned from clinical trials (16). Simultaneous delivery of large (IV bolus) doses of 5 fluorouracil with irradiation is associated with improved survival compared to treatment with radiation alone, but at a price of increased normal tissue toxicity. These side effects can be ameliorated by using protracted venous infusion. This is an efficacious approach, with a wide therapeutic index, which permits concurrent treatment of micrometastatic disease and radiation sensitization.

Combined modality therapy, including irradiation and concurrently administered 5FU based chemotherapy, has become the mainstay of therapy for anal and rectal cancers. Protracted venous infusion chemoradiation is also used in the preoperative management of rectal cancer and in the nonoperative management of anal cancers. The Gastrointestinal Tumor Study Group (GITSG) has demonstrated a significant survival advantage for patients who receive adjuvant combined radiation and bolus 5FU following curative resection of pancreatic cancer (17,18). Similar advantages have been demonstrated in unresectable pancreatic cancers. Significant advantages have also been shown for concurrent chemotherapy regiments containing 5FU in esophageal cancer (19), squamous cell carcinoma of the Head and Neck (20,21), and carcinoma of the cervix (22).

There is very limited experience with the use of capecitabine and radiation. Based on its relative selectivity and the increase in tumor cell 5FU levels, it should be expected that capecitabine will provide superior radiosensitization at equivalent or reduced systemic toxicity levels. Interestingly, it has been recently reported that radiation induces thymidine phosphorylase and enhances the efficacy of capecitabine in human cancer xenografts (23). This may further enhance the synergistic effects, and consequently the therapeutic ratio.

In RTOG study a substantial number of patients with gastrointestinal malignancies treated with concurrent radiotherapy and capecitabine at a dose of 1600 mg/m2/day (5 days a week) with very little toxicity(24 ).In phase II study of chemoradiation for rectal cancer 1650mg/m2/d of capecitabine for 14 days was safe and well-tolerated treatment(25).

In this study we will investigate the feasibility of concurrent Capecitabine and external beam radiotherapy, as well as collect preliminary data regarding the efficacy of this regimen.

OBJECTIVES

Hypothesis: Given the hypothesis that regimens employing greater intensity radiation yield higher rates of pain relief, radiosensitization using a tumor targeted drug like Xeloda should improve the rate of complete pain relief as compared to radiosensitization with 5FU alone.

Primary Objective:

To determine the frequency and duration of pain relief and narcotic relief for the proposed regimen.

Secondary Objective:

To determine the toxicity of concurrent Capecitabine and radiotherapy in breast cancer patients with bone metastases.

Eligibility Criteria

Patients with metastatic breast will be allowed on the study regardless of their prior exposure to chemotherapy. Today, there is no evidence to suggest crossresistance between radiotherapy and prior chemotherapy, or that response to radiotherapy is related in any way to the number of lines of chemotherapy used in a particular patient. Good palliative responses can often be achieved in heavily pretreated patients.

1. The patient must be 18 years of age or older.
2. The patient must have histologically proven breast adenocarcinoma.
3. Radiographic evidence of bone metastasis is required .Acceptable studies include plain radiographs, radionuclide bone scans, computed tomography scans and magnetic resonance imaging.

4 .The patient must have pain that appears to be related to the radiographically documented metastasis.

5. Patients receiving systemic therapy with Capecitabine to metastatic disease (according to health basket ).

6. Patients must have an estimated life expectancy of 3 months or greater.

7. Patients will be eligible for treatment of multiple metastases only if these can be included in no more than two treatment sites.

8. Signed study specific informed consent.

9 Karnofsky Performance Status > 40.

10. Calculated Creatinine Clearance > 50 ml/min

11.ALT and AST no greater than 3 5 times the institutional normal; bilirubin and serum creatinine no greater than 1.5 times normal; ANC greater than 1500, and platelets at least 100,00.

Exclusion Criteria

1. Prior radiation therapy or prior palliative surgery to the painful site.
2. Impending fracture of the treatment site or planned surgical fixation of the bone.
3. Patients with clinical or radiographic evidence of spinal cord or cauda equina compression.
4. Patients receiving systemic radionuclides (strontium, samarium, etc.) within 60 days prior to registration.

   PRETREATMENT EVALUATION

1. Histologic diagnosis of the primary site. 2. Radiographic assessment, with must include plain x-ray of the index lesion (s) and a bone scane.

3. Pain assessment score (BPI ). 4. Laboratory studis within 2 weeks of registration (CBC, serum ALT, AST ,total bilirubin and creatinine).

RADIATION THERAPY

1. Treatment must be given using 6-15MV photons or 6-18 MeV electrons .
2. All fields must be treated each day. Treatment volume will include the radiographic abnormality with at least a 2 cm margin. Treatment of the entire bone is not required.
3. Anterior and posterior parallel opposed fields will be used for lumbar spine, sacrum, and extremity sites. Equal weighting is recommended, although unequal weighting may be used for the lumbar or sacral spine with a ratio of doses of 1:2 AP:PA. Dose will be prescribed at mid depth at the central axis, or at the center of target volume if unequal weighting is used.

   Alternatively, the lumbar spine may be treated with a single PA field, with the dose prescribed to the mid vertebral body as defined by a lateral simulator film.
4. Single posterior fields will be used for the thoracic spine and scapula .The treatment depth is set at the middle of the vertebral body, as determined by a lateral simulation film.
5. The cervical spine may be treated with either parallel opposed lateral fields or with a single posterior field. When lateral fields are used, the isocenter should be at mid thickness, with the dose prescribed to the mid vertebral body.
6. Pubic. bone lesions will be treated with a single anterior field at a depth determined by lateral radiograph or CT scan.
7. Clavicular lesions will be treated with a single anterior field at a depth of 3 cm. The dose will be prescribed to the 3 cm depth. An alternative depth may be used as determined by CT scan or other radiographs.
8. Rib metastases may be treated with electrons or with photons. When electrons are used, the appropriate energy should be chosen such that the entire lesion is covered by the 90% (or higher) isodose curve. The dose will be prescribed to the 100% isodose line. When photons are used, parallel opposed fields may be used, with the depth prescribed to the mid thickness. Tangential fields are strongly encouraged to avoid treatment of underlying structures. A single field may be used to cover the lesion, with the depth set at the estimated depth of the rib lesion, and the dose prescribed to that level.
9. When more than one osseous site is to be included into a treatment field, the treating radiation oncologist may use different field arrangements at herlhis discretion, with the goal of providing relatively uniform coverage of the target sites and minimum inclusion of uninvolved tissues.

Radiation Dose

All patients will receive radiotherapy to a dose 30 Gy in 10fractions (3 Gy per fraction) over two weeks.

CHEMOTHERAPY

Chemotherapy with capecitabine tablets will be given concurrently with radiotherapy in the dose 1400 mg/m2 orally, in two daily divided doses.

Total daily dose rounded to the nearest 500 mg and divided into morning and evening

Doses, as per the following table:

Number of 500 mg tablets to be taken Surface Area Total Daily Dose morning evening (m2) (mg)* <= 1.08 1000 1 1 1.09 1.4 1500 2 1 1.41 1.71 2000 2 2 1.72 2.02 2500 3 2

*Total Daily Dose rounded to the nearest 500 mg and divided into morning and evening doses.

Dose Limiting Toxicity

i) >grade 3 non hematologic toxicity, except for diarrhea, nausea, vomiting, fatigue, anorexia, alopecia, fever and/or local reactions.

ii) grade 4 diarrhea lasting >3 days which is not controllable with loperamide or other such medications. Or grade 4 diarrhea that requires IV hydration.

iii) grade 4 neutropenia lasting >3 days

iv) grade 4 thrombocytopenia

v) grade 2 hand foot syndrome. Dose adjustments will be as per the following table:

Toxicity NCI Grades During a Course of Therapy Grade 1 Maintain dose Grade 2 1st appearance (non HFS) Interrupt until resolved to grade 0 1

1st appearance of HFS Interrupt until resolved to grade 0 1, then continue at 75 % of original dose.

2nd appearance Interrupt until resolved to grade 0 1, then continue at 75 % of original dose.

3rd appearance Interrupt until resolved to grade 0 1, then continue at 50 % of original dose.

4th appearance Discontinue treatment permanently Grade 3

1. st appearance Interrupt until resolved to grade 0 1, then continue at 75 % of original dose with prophylaxis where possible.
2. nd appearance Interrupt until resolved to grade 0 1, then continue at 50 % of original dose.
3. rd appearance Discontinue treatment permanently Grade 4

1st appearance Discontinue permanently or If physician deems it to be in the patient's best interest to continue, interrupt until resolved to grade 0 1, then continue at 50 % of original dose .

Dosage modifications are not recommended for grade 1 events. Therapy with capecitabine should be interrupted upon the occurrence of a grade 2 or 3 adverse experience. Once the adverse event has resolved or decreased in intensity to grade 1, then therapy may be restarted at full dose or as adjusted according to the above table. If a grade 4 experience occurs, therapy should be discontinued or interrupted until resolved or decreased to grade 1, and therapy should be restarted at 50% of the original dose. Doses of capecitabine omitted for toxicity are not replaced or restored; instead the patient should resume the planned treatment cycles. Once the dose has been reduced it should not be increased at a later time.

Toxicity

CAPECITABINE can induce diarrhea, sometimes severe. Patients with severe diarrhea should be carefully monitored and given fluid and electrolyte replacement if they become dehydrated. National Cancer Institute of Canada (NCIC grade 2 diarrhea is defined as an increase of 4 to 6 stools/day or nocturnal stools, grade 3 diarrhea as an increase of 7 to 9 stools/day or incontinence and malabsorption, and grade 4 diarrhea as an increase of >10 stools/day or grossly bloody diarrhea or the need for parenteral support. If grade 2, 3 or 4 diarrhea occurs, administration of capecitabine should be immediately interrupted until the diarrhea resolves or decreases in intensity to grade 1. Following grade 3 or 4 diarrhea, subsequent doses of capecitabine should be decreased. Standard antidiarrheal treatments (eg, loperamide) are recommended. Necrotizing enterocolitis (typhlitis) has also been reported.

Hand and foot syndrome (palmar plantar erythrodysesthesia or chemotherapy induced acral erythema) is characterized by the following: numbness, dysesthesia/paresthesia, tingling, painless or painful swelling, erythema, desquamation, blistering and severe pain. Grade 2 hand and foot syndrome is defined as painful erythema and swelling of the hands and/or feet and/or discomfort affecting the patient's activities of daily living. Grade 3 hand and¬foot syndrome is defined as moist desquamation, ulceration, blistering and severe pain of the hands and/or feet and/or severe discomfort that causes the patient to be unable to work or perform activities of daily living. If grade 2 or 3 hand and foot syndrome occurs, administration of capecitabine should be interrupted until the event resolves or decreases in intensity to grade 1. Following the occurrence of grade 2 handand foot syndrome, subsequent doses of capecitabine should be decreased.

There has been cardiotoxicity associated with fluorinated pyrimidine therapy, including myocardial infarction, angina, dysrhythmias, cardiogenic shock, sudden death and electrocardiograph changes. These adverse events may be more common in patients with a prior history of coronary artery disease.

Patients with mild to moderate hepatic dysfunction due to liver metastases should be carefully monitored when capecitabine is administered. The effect of severe hepatic dysfunction on the disposition of capecitabine is not known. If drug related grade 2 4 elevations in bilirubin occur, administration of capecitabine should be immediately interrupted until the hyperbilirubinernia resolves or decreases in intensity to grade 1. NCIC grade 2 hyperbilirubinernia is defined as 1.5 x normal, grade 3 hyperbilirubinemia as 1.5 3 x normal and grade 4 hyperbilirubinemia as >3 x normal.

Increases in adverse events have been noted in patients with reduced renal function. Therefore, patients will be excluded for a calculated creatinine clearance of less than 50 ml/min.

Myelosuppression was rare.

Assessment of Response

Pain scores and narcotic scores will be determined using the guidelines in following table:

PAIN AND NARCOTIC CATEGORIES AND SCORES PAIN ANALGESIA Severity 0 No pain 0 None I Mild I Analgesics (ASA, Bufferin, Tylenol, Anacin, etc.) 2 Moderate 2 Mild Narcotic, (< 112 gr. codeine, Darvon, etc.) 3 Severe 3 Moderate Narcotic (> 112 < gr. codeine, Percoan, etc) 4 Strong 4 Narcotic, (> 1 gr. codeine, demerol, morphine, etc) Frequency 0 None 0 None I Occasional (< daily) I p.r.n. (< daily) 2 Intermittent (at least daily) 2 q.d. (I tab. or cap./day) 3 Frequent (>. I < 3 daily) 3 b.i.d. t.i.d. (> I < 4 tab. or cap./day) 4 Constant (most of the time) 4 > t.i.d. (> 4 tab. or cap./day)

Pain Score = Pain Severity Grade x Pain Frequency Grade Narcotic Score = Analgesia Severity Grade x Analgesic Frequency Grade

Response will be evaluated by questionnaires at follow up visit at 2, 4 and 8 weeks after completion of radiotherapy and by phone call interviews (when necessary for completeness) in poor compliance patients.

The "worst pain score" will be used as response endpoint. The time to maximal pain relief is the time from the first day of irradiation to the time of the lowest pain score for average pain.

Response Definitions

Complete response is defined as an average pain score of 0 for two consecutive analysis periods. Narcotic consumption must not be increased. Partial response. A decrease of at least 2 points in the worst pain score for two consecutive analysis periods. Narcotic consumption must not be increased. No response (any of the following): A pain score that does not change within 8 weeks from the start of radiation therapy.

A 2 point increase in worst pain score that is sustained at a higher level in the month following the first day of radiation therapy.

A pain score that drops by at least 2 points and subsequent sustained rise (on 2 successive questionnaires) of pain score by at least 2 points. Any patient with progressive pain in the treated area should have plain radiographs of the area to assess for bone stability and pathologic fracture.

References.

1.

Hoskin PJ. Scientific and clinical aspects of radiotherapy in the relief of bone pain. Cancer Surv. 7:69, 1988.

2. Tong D, Gillick L, Hendrickson FR. The palliation of symptomatic osseous metastases: the

results of the Radiation Therapy Oncology Group. Cancer 1982; 50: 893.

3. Hoskin PJ, Price P, Easton D, et a]. A prospective randomized trial of 4 Gy or 8 Gy single doses

in the treatment of metastatic bone pain. Radiotherapy and Oncology 23:74 78, 1992.

4. Price P, Hoskin PJ, Easton D, et al. Prospective randomized trial of single and multifraction

radiotherapy schedules in the treatment of painful bony metastases. Radiotherapy and Oncology 6: 247 255, 1986.

Okawa T, Kita M, Goto M, et al. Randomized prospective clinical study of small, large and twice a day fraction radiotherapy for painful bone metastases. Radiotherapy and Oncology 13: 99 104, 1988.

6. Madsen EL, Painful bone metastases: Efficacy of radiotherapy assessed by the patients: A

randomized trial comparing 4 Gy x 6 versus 10 Gy x 2. Int. J. Radiat. Oncol. Biol. Phys. 9:1775¬ 1779, 1983.

7. Blitzer PH. Reanalysis of the RTOG study of the palliation of symptomatic osseous metastasis.

Cancer 1985; 55: 1468 1472.

8. Orton CG, Ellis F, A simplification in the use of the NSD concept in practical radiotherapy. Br.

J. Radiol. 1973; 46:529 537.

9. Daut R, Cleeland C, Flanery R: Development of the Wisconsin Brief Pain questionnaire to assess

pain in cancer and other diseases. Pain 17:197 210, 1983.

10.

11.

12.

13.

14.

Cella DF, Tulsky DS, Gray G, et al.: The Functional Assessment of Cancer Therapy Scale: Development and validation of the general measure. J Clin Oncol 11:570 579, 1993.

Ben Josef E, Shamsa F, Youssef E, Porter AT. External beam radiotherapy for painful osseous metastases: pooled data dose response analysis. Int J Radiat Oncol Biol Phys 45(3):715 719, 1999.

Byfield JE, calabro Jones P, Klisak 1, et al. Pharmacologic requirements for obtaining sensitization of human tumor cells in vitro to combined r fluorouracil or ftorafur and x rays. Int J Radiat Oncol Biol Phys 1982, 8:1923 33.

Nakajima V, Miyamoto Y, Tanabe M, et al. Enhancement of mammalian cell killing by 5fluorouracil in combination with x rays. Cancer Res 39:3763 3767, 1979.

Lawrence TS, Davis MA, Maybaum I Dependence of 5 fluorouracil mediated radiosensitization on DNA directed effects. Int J Radiat Oncol Biol Phys 1994, 29(3):519 23.

15. Weinberg MJ, Rauth AM. 5 fluorouracil infusion and fractionated doses of radiation: Studies with a murine sqamous cell carcinoma. Int J Radiat Oncol Biol Phys 13: 1691 1699, 1987.

Rich TA. Infusional chemoradiation for rectal and anal cancers. Oncology (Huntingt) 1999, 13(10 Suppl 5):131 4.

17. Gastrointestinal Tumor Study Group. Further evidence of effective adjuvant combined radiation and chemotherapy following curative resection of pancreatic cancer. Cancer 1987, 59(12):2006¬ 10.

18. Kalser MH, Ellenberg SS. Pancreatic cancer. Adjuvant combined radiation and chemotherapy following curative resection. Arch Surg 1985, 120(8):899 903.

19. al Sarraf M, Martz K, Herskovic A, Leichman L, Brindle JS, Vaitkevicius VK, Cooper J, Byhardt R, Davis L, Emami B. Progress report of combined chemoradiotherapy versus radiotherapy alone in patients with esophageal cancer: an intergroup study. J Clin Oncol 1997, 15(l):277 84.

20. Wendt TG, Grabenbauer GG, Rodel CM, Thiel HJ, Aydin H, Rohloff R, Wustrow TP, Iro H, Popella C, Schalhorn A. Simultaneous radiochemotherapy versus radiotherapy alone in advanced head and neck cancer: a randomized multicenter study. J Clin Oncol 1998, 16(4):1318 24.

21. Al Sarraf M, LeBlanc M, Giri PG, Fu KK, Cooper J, Vuong T, Forastiere AA, Adams G, Sakr WA, Schuller DE, Ensley JF. Chemoradiotherapy versus radiotherapy in patients with advanced nasopharyngeal cancer: phase III randomized Intergroup study 0099. J Clin Oncol 1998, 16(4):1310 7.

22. Morris M, Eifel PJ, Lu J, Grigsby PW, Levenback C, Stevens RE, Rotman M, Gershenson DM, Mutch DG. Pelvic radiation with concurrent chemotherapy compared with pelvic and para aortic radiation for high risk cervical cancer. N Engl J Med 1999, 340(15):1137 43.

23. Sawada N, Ishikawa T, Sekiguchi F, Tanaka Y, Ishitsuka H. X ray irradiation induces thymidine phosphorylase and enhances the efficacy of capecitabine in human cancer xenografts. Clin Cancer Res 1999, 5(10):2948 53.

24. U.N.Vaishampayan, E. Ben-Josef, P.A. Philip, V.K. Vaitkevicius, K.J. Levin and A.F. Shields. A single- institution experience with concurrent capecitabine and radiation therapy in gastrointestinal malignancies . Int J Radiat Oncol Biol Phys ,2002, 53,675-679.

25. Jun-Sang Kim, Jae-Sung Kim, Moon-June Cho and Wan-Hee Yoon .Preoperative chemoradiation using oral capecitabine in locally advanced rectal cancer. Int J Radiat Oncol Biol Phys ,2002,54,403-408.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be 18 years of age or older
2. The patient must have histologically proven breast adenocarcinoma
3. Radiographic evidence of bone metastasis is required .Acceptable studies include plain radiographs, radionuclide bone scans, computed tomography scans and magnetic resonance imaging
4. The patient must have pain that appears to be related to the radiographically documented metastasis
5. Patients receiving systemic therapy with Capecitabine to metastatic disease (according to health basket)
6. Patients must have an estimated life expectancy of 3 months or greater
7. Patients will be eligible for treatment of multiple metastases only if these can be included in no more than two treatment sites
8. Signed study specific informed consent
9. Karnofsky Performance Status > 40
10. Calculated Creatinine Clearance > 50 ml/min
11. ALT and AST no greater than 3 5 times the institutional normal; bilirubin and serum creatinine no greater than 1.5 times normal; ANC greater than 1500, and platelets at least 100,00

Exclusion Criteria:

1. Prior radiation therapy or prior palliative surgery to the painful site
2. Impending fracture of the treatment site or planned surgical fixation of the bone
3. Patients with clinical or radiographic evidence of spinal cord or cauda equina compression
4. Patients receiving systemic radionuclides (strontium, samarium, etc.) within 60 days prior to registration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2004-05; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in pain score at 12 wks | 12 weeks
  Patients were asked to score their pain on a scale of 0 (no pain) to 10 (worst possible pain) before treatment and at 1, 2, 4, 8 and 12 weeks after treatment initiation.

SECONDARY OUTCOMES:
Change in pain medications consupmtion at 12 weeks compared to basline | 12 weeks
  Consumption of analgesics was evaluated by the physician using the 5-point WHO score, as follows: level 0, no analgesics required; level 1, non-narcotic analgesics required occasionally; level 2, non-narcotic analgesics required regularly; level 3, narcotic analgesics required occasionally; level 4, narcotic analgesics required regularly

CONTACTS AND LOCATIONS:
Overall Officials: Yulia Kundel, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Beilinson Campus, Petah Tikva, Israel

REFERENCES:
- [Derived] Kundel Y, Nasser NJ, Purim O, Yerushalmi R, Fenig E, Pfeffer RM, Stemmer SM, Rizel S, Symon Z, Kaufman B, Sulkes A, Brenner B. Phase II study of concurrent capecitabine and external beam radiotherapy for pain control of bone metastases of breast cancer origin. PLoS One. 2013 Jul 10;8(7):e68327. doi: 10.1371/journal.pone.0068327. Print 2013. PMID 23874586